CLINICAL TRIAL: NCT04170634
Title: Tumoral Bone Strength Assessment by Numerical Simulation Using Quantitative CT (Computed Tomography) : the MEKANOS Study
Brief Title: Tumoral Bone Strength Assessment by Numerical Simulation Using Quantitative CT : the MEKANOS Study
Acronym: MEKANOS
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0642
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Metastases to Bone; Metastatic Breast Cancer; Metastatic NSCLC
Keywords: osteolytic secondary tumoral lesion; femur; vertebrae; qCT routine imagery
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood collection: 12 mL of blood (4 mL for plasma and 8 mL for serum isolation) will be collected at the baseline, concomitantly to routine blood analysis. Plasma and serum will be stored at -80°C for further analysis on bone markers (CTX: C-Terminal Telopeptide, DKK1: Dickkopf-1, ALP: Alkaline Phosphatase and P1NP: Procollagen I N-Terminal Propeptide).
  Ancillary study: The ancillary study will allow the experimental characterization of the mechanical properties of the bone and soft tissue tumor volume, in order to integrate them into the simulation and conduct a sensitivity study for a wide range of values
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with bone metastases at risk of fracture: Adult patients with tumor osteolytic bone lesions located in proximal femur and/or vertebrae secondary to a myeloma or a breast, lung (NSCL: Non-Small Cell Lung), bladder, thyroid or kidney cancer. The target vertebrae or femur has to be naïve of localized treatment (interventional radiology - cementoplasty, cryotherapy, radiofrequency…). Previous exposure to systemic oncological treatments (chemotherapy, targeted therapy, immunotherapy…) and bone treatments are allowed if administered for less than 3 months.
  Interventions: Other: Evaluation of the fracture risk using data from routine qCT (quantitative Computed Tomography) scan and numerical simulation

INTERVENTIONS:
Other: Evaluation of the fracture risk using data from routine qCT (quantitative Computed Tomography) scan and numerical simulation — Assessment of the mechanical tumor bone strength by numerical simulation using qCT routine imagery of proximal femur (applying a monopodal standing load) and vertebrae (applying a uniaxial compression load).

SUMMARY:
Osteolytic bone metastases and myeloma bone lesions are responsible of long bone and vertebral fractures leading to restricted mobility, surgery and medullar compression that severely alter quality of life and that have a huge medico-economic impact. It has been estimated that 50% of the patients with bone metastasis will encounter bone complications. In the recent years, Bone Oncology Multidisciplinary Meetings have been developed to optimize bone metastases management for each patient in harmony with oncology program.

The assessment of the fracture risk of bone metastasis remains fairly empirical and is based on simple radiography. The Mirel's score for long bones is focused on the extent of cortical defect caused by bone metastasis to identify high-risk patients at risk of fracture during surgery. It is old, little used in routine and lacks sensitivity and specificity. The SINS (Spinal Instability Neoplastic Score) score is the reference for vertebrae. Today, most patients with fracture-risk bone metastasis benefit from a lesion-centered CT scan to better characterize its extent and position but the interpretation remains qualitative. Metastases are considered as an air cavity and the mechanical properties of the tumor are not evaluated. However, many other parameters from the CTscan are available such as cortical or trabecular compartment densitometry, cortical thickness, tumor volume, and position of lysis in the bone.

Based on experience acquired by the service in the evaluation of bone mechanical strength on benign bones, the investigator aim at integrating in the numerical simulation the mechanical properties of both bone and tumor, in order to evaluate the mechanical strength of the pathological bone using a numerical simulation model (finite element analysis-FEA).

MEKANOS will enroll patients with bone metastases of breast, lung, kidney, thyroid or bladder cancer and myeloma lesions affecting the vertebrae or the upper end of the femur.

The resistance obtained will be compared to that of an intact bone. The best predictive parameters of mechanical strength (position of lysis, tumor nature, and bone architecture) will be then determined. Finally, the added value of this technique in relation to historical fragility scores (Mirel's and SINS scores) will be assessed.

The ultimate goal is to provide tools to assess fracture risk and improve the preventive management of bone metastases in harmony with the referring oncologist

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years of age).
* Patients who do not object to participating in the study. For patients participating to the biological collection: signature of the written informed consent..
* Patients with secondary tumor lesion(s) of mammary or pulmonary non-small cell, renal, bladder, thyroid or myeloma bone origin.
* Existence of a CT scan focused on the target lesion (or which will be performed as part of the care), performed within a time window of 30 days before and 20 days after inclusion, as part of the patient's usual bone management.
* Target location: upper end of the femur (1/3 proximal) and/or vertebrae. Several locations are possible for the same patient, provided that the inclusion criteria are met for each target.
* Size of target lesion: either diffuse permeative or > 15 mm in size.
* Exposure to systemic bone therapy for 3 months or less (daily clodronate or denosumab, zoledronic acid, monthly pamidronate) is allowed
* Patients who received previous systemic oncological treatments (chemotherapy, targeted therapy, immunotherapy…) are eligible.

Exclusion Criteria:

* Patients who have received targeted treatment at the target location either in the form of radiotherapy, surgery or interventional radiology (cementoplasty, cryotherapy, radiofrequency).
* Fractured pathological target bone.
* For the femur target, the patient must not have a hip prosthesis on either side (target or contralateral)
* Patients under trusteeship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with predominantly osteolytic tumor involvement related either to myeloma or bone metastases of lung, breast, bladder, thyroid or kidney cancer.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2019-11-28 (Actual); Primary Completion 2026-11-28 (Estimated); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
Measurement of mechanical strength of tumor proximal femur or tumor vertebrae obtained by numerical simulation using the finite element analysis (FEA) method. | 24 months
  Measurement of mechanical strength (expressed in Newton : N), monopodal support at the upper end of the femur and uniaxial compression on the vertebrae, obtained by numerical simulation using the finite element analysis (FEA) method.
  As an indication, the average resistance of a femur of an elderly patient in monopod support is on average 9000 N and that of the L3 vertebra in uniaxial compression is on average 2700 N.
  Comparative values will also be obtained on the healthy contralateral femur and an adjacent healthy vertebra of each patient

CONTACTS AND LOCATIONS:
Overall Officials: Cyrille CONFAVREUX, PR, Principal Investigator — Service de Rhumatologie
Locations (12):
- France (12):
  - Service de rhumatologie, CHU d'Angers, Angers
  - Ch Annecy Genevois, Annecy
  - Service de radiothérapie, Institut Jean-Perrin, Clermont-Ferrand
  - Service de rhumatologie, CH Annemasse, Contamine-sur-Arve
  - Service d'onco-rhumatologie, Centre Oscar Lombret, Lille
  - Service de Radiothérapie, Centre Léon Bérard, 28 Prom. Léa et Napoléon Bullukian, Lyon
  - Service d'oncologie médicale, Institut Curie, 26 rue d'Ulm, Paris
  - Service de Radiologie, Hôpital Cochin, Assistance Publique - Hôpitaux de Paris, Paris
  - Service de Rhumatologie, Hospices Civils de Lyon, Groupement Hospitalier Lyon Sud, Pierre-Bénite
  - Service de rhumatologie, CHU de Poitiers, Poitiers
  - Service de rhumatologie, CHU de Saint Etienne, Saint-Priest-en-Jarez
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy